CLINICAL TRIAL: NCT02113449
Title: A Study to Assess the Market Potential of a Carbon Dioxide Nasal Spray in Congested Subjects
Brief Title: Market Potential of Carbon Dioxide Nasal Spray
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202181; RH01910 (Other: GSK)
Record Dates: First submitted 2014-02-06; First posted 2014-04-14 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Nasal Congestion
Keywords: Carbon Dioxide, Allergy symptoms
MeSH Terms: conditions — Nasal Obstruction | interventions — Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Participants will receive one dose of nasal carbon dioxide (CO2) in the study clinic under medical supervision, followed by an additional six days of at home use, up to 4 times per day.
  Interventions: Drug: Carbon Dioxide

INTERVENTIONS:
Drug: Carbon Dioxide — Nasal administration of carbon dioxide (CO2) through the delivery device for 10 seconds

SUMMARY:
Carbon dioxide (CO2) is a naturally occurring gas that readily diffuses across body tissues and membranes. Data from earlier clinical studies conducted in 975 subjects with allergic rhinitis have shown that nasally administered CO2 may provide relief of the associated symptoms. Symptom relief has been shown to occur as soon as 10 minutes after administration, and may persist for four to six hours.

This study aims to assess the consumer appeal of a prototype CO2 delivery device, as well as evaluate its perceived effectiveness for nasal congestion. Properly consented subjects who qualify and choose to participate in the clinical study will be administered nasal CO2 under medical supervision, wait a period of 1 hour in clinic, and then be dispensed a device for self-treatment at home. Subjects will return to the clinic on day 7 for final evaluation and completion of assessment questionnaires.

DETAILED DESCRIPTION:
This study will be conducted in two parts. In the first part of the study, recruited subjects with nasal congestion will view a description of a new treatment option (concept). Interested subjects will be offered the opportunity to enter the clinical trial. Subjects who consent and are found otherwise eligible will then receive one dose of CO2 in the study clinic under medical supervision. Afterward, subjects who wish to continue will be allowed to take the administration device home for an additional six days of use (study part 2).

During the at-home use portion of the study, subjects will use a diary to record the number of times the product was used and their nasal congestion symptoms before and after use.

At the end of the study period, subjects will return to the study center for global assessment of their impressions of treatment and to answer questions designed to estimate market acceptability. Subjects may be asked to participate voluntarily in a market research focus group following their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participant who demonstrate understanding of, and willingness to participate in the study
* Aged at least 18 years.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee
* Participant has perception of Nasal Breathing score ≤70 mm (Visual Analogue Scale) on the evaluation day
* Females of childbearing potential who are, in the opinion of the investigator, practising a reliable method of contraception.

Exclusion Criteria:

* Women who are known to be pregnant or who have a positive pregnancy test, or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Recent history (within the last 2 years) of alcohol or other substance abuse.
* Medical history of significant respiratory impairment.
* No history of product purchase for treatment of nasal congestion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - Radiant Research - Chandler, AZ, Chandler, Arizona
  - Radiant Research - Pinellas Park, FL, Pinellas Park, Florida
  - TKL Research Inc, Paramus, New Jersey
  - Radiant Research - Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Johnson SM, Hamilton AM, Lauersen LA. A phase IV, single-center, crossover evaluation of the efficacy of an external nasal dilator strip in children with nasal congestion. Allergy Asthma Proc. 2016 May;37(3):242-7. doi: 10.2500/aap.2016.37.3950. PMID 27178892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult subjects with nasal congestion were recruited at the study sites from their volunteer database and through advertising.
Pre-assignment Details: This was a 2-part study. In Part 1, recruited participants viewed a description of new treatment option (concept). Interested participants entered the trial. Eligible participants who consented received one dose of nasal CO2 in the clinic under medical supervision. Participants who wished to continue took the device home for 6 days (Part 2).
Groups:
- CO2 Nasal Spray: CO2 spray was administered for 10 seconds per nostril. Participants received one dose of nasal CO2 in the study clinic under medical supervision, followed by an additional six days of at home use, up to 4 times per day
Period: Overall Study
Arm/Group | CO2 Nasal Spray
Started | 147
Completed | 143
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Which One Product That Relieves Nasal Congestion do You Buy Most Often?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked as part of screening survey prior to concept viewing. If the participant answered "I do not purchase any product to relieve congestion" the participant was excluded. Participants could select only one option available.
Time Frame: 7 days
Population: The per protocol (PP) population was the primary population for analysis. Of the 143 participants who completed this study, 10 participants had device failure (device that didnot perform well), and therefore 133 participants were included in PP population.
Measure: Number; unit: Participants
Groups:
- All Participants: The participants were asked in the beginning which medication they purchase to relieve nasal congestion. Participant could select only one option available. If the participant answered "I do not purchase any product to relieve congestion" the participant was excluded. Participants could select only one option available.
Arm/Group | All Participants
Number analyzed (Participants) | 133
Participants
  Allergy medications | 46
  Medicated nasal sprays | 29
  Nasal rinses | 6
  Nasal strips | 3
  Non-medicated/saline nasal sprays/gels | 14
  Non-medicinal remedies | 6
  Sinus/cold medications | 15
  Prescription nasal sprays/inhalers | 14
  Prescription allergy medications | 0

2. Primary Outcome: Which of the Statements Best Describes the Extent to Which the Spray Reached Your Expectations?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked after the first use. Participants could select only one option.
Time Frame: 7 days
Population: The per protocol (PP) population was the primary population for analysis. Of the 143 participants who completed this study, 10 participants had device failure (device that did not perform well), and therefore 133 participants were included in PP population.
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Much better than you expected | 45
  A little better than you expected | 48
  Just as you expected | 27
  Not as good as you expected | 9
  Not nearly as good as you expected | 4

3. Primary Outcome: If the Product You Just Tried (After First Dose) Was Available for the Following Price: $12.99 for 40 Doses, How Likely Would You be to Buy it?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked after the first dose of the product. Participants could select only one option.
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Definitely would buy | 29
  Probably would buy | 50
  Might or might not buy | 40
  Probably would not buy | 9
  Definitely would not buy | 5

4. Primary Outcome: Would You be Interested in Taking the Spray Product Home and Using it Over the Next Week?
Description: as for outcome 3
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Yes | 133
  No | 0

5. Primary Outcome: Which of the Following Statements Best Describes the Extent to Which the Spray Reached Your Expectations?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked after at-home use of the product. Participants could select only one option.
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Much better than your usual product | 43
  A little better | 35
  As good | 22
  Not quite as good | 16
  Not nearly as good | 17

6. Primary Outcome: Divide 11 Points Between Two Products (CO2 Nasal Spray and Brand Selected at Q1)?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked after at-home use of the product. Participants could select only one option. It was done to compare the spray with the product selected by the participant in Q1. There were 11 points between the two products that participants could divide anyways thet wanted (11-0, 10-1, 9-2, 8-3, 7-4 or 6-5 etc). The more the participant liked a product compared to other, the higher the number of points were to be given to that product.
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- C02 Nasal Spray: CO2 spray was administered for 10 seconds per nostril. Participants received one dose of nasal CO2 in the study clinic under medical supervision, followed by an additional six days of at home use, up to 4 times per day
Arm/Group | C02 Nasal Spray
Number analyzed (Participants) | 133
Participants
  0 for CO2 Nasal Spray | 12
  1 for CO2 Nasal Spray | 4
  2 for CO2 Nasal Spray | 5
  3 for CO2 Nasal Spray | 5
  4 for CO2 Nasal Spray | 13
  5 for CO2 Nasal Spray | 13
  6 for CO2 Nasal Spray | 26
  7 for CO2 Nasal Spray | 19
  8 for CO2 Nasal Spray | 13
  9 for CO2 Nasal Spray | 11
  10 for CO2 Nasal Spray | 6
  11 for CO2 Nasal Spray | 6

7. Primary Outcome: If the Product You Just Tried (After At-home Use) Was Available for the Following Price: $12.99 for 40 Doses, How Likely Would You be to Buy it?
Description: as for outcome 5
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Definitely would buy | 40
  Probably would buy | 38
  Might or might not buy | 21
  Probably would not buy | 18
  Definitely would not buy | 16

8. Primary Outcome: How Many Packages Would You Buy?
Description: There was one questionnaire used in this study which was divided into 3 parts: screening survey, after product trial questions, and at home usage experience.This question was asked after at-home use of the product. Participants could select only one option.
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  1 | 54
  2 | 20
  3 | 6
  4 | 1
  5 | 1
  Missing | 51

9. Primary Outcome: Which One Statement Best Describes How Often, if Ever, You Think You Would Buy the Spray Product in the Future?
Description: There was one questionnaire used in this study which is divided into 3 parts: screening survey, after product trial questions, and at home usage experience. This question was asked after at-home use of the product. Participants could select only one option.
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  More than once a week | 43
  Once a week | 2
  Once every 2 weeks | 16
  Once every 3 weeks | 9
  Once a month | 30
  Once every 6 weeks | 10
  Once every 2 months | 12
  Once every 3 months | 7
  Once every 4-5 months | 4

10. Primary Outcome: How Often do You Think This Spray Product Would Last for You Personally?
Description: as for outcome 9
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  1 Week | 2
  2 Weeks | 17
  3 Weeks | 17
  1 Month | 28
  6 Weeks | 15
  2 Months | 10
  3 Months | 4
  4-5 Months | 3
  6 Months | 3
  9 Months | 1
  1 Year | 6
  More than 1 year | 3
  Missing | 24

11. Primary Outcome: Provide a Score From 1-7 to Some Statements, Depending on How Much You Think Each Statement Applies or Does Not Apply to the Spray Product That You Used
Description: A score of 1 indicates that the statement does not apply at all to the product that you used. A score of 7 indicates that it applies completely to it. You can use any score from 1 to 7 to indicate how much or how little you think the statement applies to this product
Time Frame: 7 days
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- CO2 Nasal Spray: Score from 1 to 7 indicates how much or how little you think the statement applies to this product. A score of 1 indicates that the statement does not apply at all to the product that you used. A score of 7 indicates that it applies completely to it
Arm/Group | CO2 Nasal Spray
Number analyzed (Participants) | 133
Participants
  Is easy to use; 1 | 2
  Is easy to use; 2 | 2
  Is easy to use; 3 | 5
  Is easy to use; 4 | 5
  Is easy to use; 5 | 22
  Is easy to use; 6 | 15
  Is easy to use; 7 | 82
  Provides effective relief for nasal congestion; 1 | 10
  Provides effective relief for nasal congestion; 2 | 7
  Provides effective relief for nasal congestion; 3 | 10
  Provides effective relief for nasal congestion; 4 | 11
  Provides effective relief for nasal congestion; 5 | 21
  Provides effective relief for nasal congestion; 6 | 21
  Provides effective relief for nasal congestion; 7 | 53
  Provides instant relief; 1 | 13
  Provides instant relief; 2 | 7
  Provides instant relief; 3 | 8
  Provides instant relief; 4 | 13
  Provides instant relief; 5 | 28
  Provides instant relief; 6 | 24
  Provides instant relief; 7 | 40
  Provides long lasting relief; 1 | 13
  Provides long lasting relief; 2 | 8
  Provides long lasting relief; 3 | 16
  Provides long lasting relief; 4 | 18
  Provides long lasting relief; 5 | 16
  Provides long lasting relief; 6 | 30
  Provides long lasting relief; 7 | 32
  Helps you breathe better; 1 | 9
  Helps you breathe better; 2 | 6
  Helps you breathe better; 3 | 7
  Helps you breathe better; 4 | 12
  Helps you breathe better; 5 | 15
  Helps you breathe better; 6 | 26
  Helps you breathe better; 7 | 58
  Drug free; 1 | 7
  Drug free; 2 | 1
  Drug free; 3 | 2
  Drug free; 4 | 5
  Drug free; 5 | 8
  Drug free; 6 | 12
  Drug free; 7 | 98
  Is a product for someone like me; 1 | 25
  Is a product for someone like me; 2 | 5
  Is a product for someone like me; 3 | 4
  Is a product for someone like me; 4 | 4
  Is a product for someone like me; 5 | 10
  Is a product for someone like me; 6 | 19
  Is a product for someone like me; 7 | 66
  Prevents allergy symptoms; 1 | 24
  Prevents allergy symptoms; 2 | 8
  Prevents allergy symptoms; 3 | 13
  Prevents allergy symptoms; 4 | 11
  Prevents allergy symptoms; 5 | 18
  Prevents allergy symptoms; 6 | 20
  Prevents allergy symptoms; 7 | 39
  Effectively treats allergy symptoms; 1 | 15
  Effectively treats allergy symptoms; 2 | 8
  Effectively treats allergy symptoms; 3 | 11
  Effectively treats allergy symptoms; 4 | 11
  Effectively treats allergy symptoms; 5 | 19
  Effectively treats allergy symptoms; 6 | 27
  Effectively treats allergy symptoms; 7 | 42
  Is a brand I trust; 1 | 19
  Is a brand I trust; 2 | 10
  Is a brand I trust; 3 | 4
  Is a brand I trust; 4 | 15
  Is a brand I trust; 5 | 17
  Is a brand I trust; 6 | 17
  Is a brand I trust; 7 | 51
  Is a good value for the money; 1 | 19
  Is a good value for the money; 2 | 5
  Is a good value for the money; 3 | 10
  Is a good value for the money; 4 | 9
  Is a good value for the money; 5 | 25
  Is a good value for the money; 6 | 23
  Is a good value for the money; 7 | 42
  Is very effective; 1 | 14
  Is very effective; 2 | 7
  Is very effective; 3 | 6
  Is very effective; 4 | 12
  Is very effective; 5 | 19
  Is very effective; 6 | 25
  Is very effective; 7 | 50
  Is safe to use every day; 1 | 15
  Is safe to use every day; 2 | 6
  Is safe to use every day; 3 | 8
  Is safe to use every day; 4 | 7
  Is safe to use every day; 5 | 12
  Is safe to use every day; 6 | 27
  Is safe to use every day; 7 | 58
  Helps you sleep better; 1 | 29
  Helps you sleep better; 2 | 7
  Helps you sleep better; 3 | 6
  Helps you sleep better; 4 | 10
  Helps you sleep better; 5 | 16
  Helps you sleep better; 6 | 17
  Helps you sleep better; 7 | 48
  Effectively treats multiple symptoms; 1 | 25
  Effectively treats multiple symptoms; 2 | 10
  Effectively treats multiple symptoms; 3 | 9
  Effectively treats multiple symptoms; 4 | 10
  Effectively treats multiple symptoms; 5 | 22
  Effectively treats multiple symptoms; 6 | 25
  Effectively treats multiple symptoms; 7 | 32
  Does not cause side effects; 1 | 17
  Does not cause side effects; 2 | 6
  Does not cause side effects; 3 | 8
  Does not cause side effects; 4 | 13
  Does not cause side effects; 5 | 15
  Does not cause side effects; 6 | 19
  Does not cause side effects; 7 | 55
  Helps you feel better the next day; 1 | 23
  Helps you feel better the next day; 2 | 9
  Helps you feel better the next day; 3 | 10
  Helps you feel better the next day; 4 | 9
  Helps you feel better the next day; 5 | 20
  Helps you feel better the next day; 6 | 24
  Helps you feel better the next day; 7 | 38
  Helps you breathe more freely; 1 | 10
  Helps you breathe more freely; 2 | 8
  Helps you breathe more freely; 3 | 6
  Helps you breathe more freely; 4 | 6
  Helps you breathe more freely; 5 | 15
  Helps you breathe more freely; 6 | 24
  Helps you breathe more freely; 7 | 64
  Does not interact with any medications; 1 | 13
  Does not interact with any medications; 2 | 1
  Does not interact with any medications; 3 | 4
  Does not interact with any medications; 4 | 5
  Does not interact with any medications; 5 | 10
  Does not interact with any medications; 6 | 21
  Does not interact with any medications; 7 | 79
  Safe to use multiple times in a day; 1 | 14
  Safe to use multiple times in a day; 2 | 9
  Safe to use multiple times in a day; 3 | 3
  Safe to use multiple times in a day; 4 | 6
  Safe to use multiple times in a day; 5 | 17
  Safe to use multiple times in a day; 6 | 17
  Safe to use multiple times in a day; 7 | 67
  Prevents the release of histamine; 1 | 23
  Prevents the release of histamine; 2 | 6
  Prevents the release of histamine; 3 | 5
  Prevents the release of histamine; 4 | 9
  Prevents the release of histamine; 5 | 16
  Prevents the release of histamine; 6 | 28
  Prevents the release of histamine; 7 | 46
  Prevents nasal congestion before it starts; 1 | 20
  Prevents nasal congestion before it starts; 2 | 11
  Prevents nasal congestion before it starts; 3 | 10
  Prevents nasal congestion before it starts; 4 | 12
  Prevents nasal congestion before it starts; 5 | 26
  Prevents nasal congestion before it starts; 6 | 22
  Prevents nasal congestion before it starts; 7 | 32
  Stops nasal congestion where it starts; 1 | 16
  Stops nasal congestion where it starts; 2 | 9
  Stops nasal congestion where it starts; 3 | 5
  Stops nasal congestion where it starts; 4 | 10
  Stops nasal congestion where it starts; 5 | 21
  Stops nasal congestion where it starts; 6 | 28
  Stops nasal congestion where it starts; 7 | 44
  Can be used with other nasal congestion remedy; 1 | 24
  Can be used with other nasal congestion remedy; 2 | 4
  Can be used with other nasal congestion remedy; 3 | 6
  Can be used with other nasal congestion remedy; 4 | 8
  Can be used with other nasal congestion remedy; 5 | 16
  Can be used with other nasal congestion remedy; 6 | 24
  Can be used with other nasal congestion remedy; 7 | 51
  Can feel it working instantly; 1 | 13
  Can feel it working instantly; 2 | 7
  Can feel it working instantly; 3 | 6
  Can feel it working instantly; 4 | 8
  Can feel it working instantly; 5 | 11
  Can feel it working instantly; 6 | 30
  Can feel it working instantly; 7 | 58
  Works like no other product; 1 | 14
  Works like no other product; 2 | 3
  Works like no other product; 3 | 7
  Works like no other product; 4 | 10
  Works like no other product; 5 | 15
  Works like no other product; 6 | 31
  Works like no other product; 7 | 53
  Relieves my symptoms instantly; 1 | 16
  Relieves my symptoms instantly; 2 | 4
  Relieves my symptoms instantly; 3 | 11
  Relieves my symptoms instantly; 4 | 10
  Relieves my symptoms instantly; 5 | 16
  Relieves my symptoms instantly; 6 | 30
  Relieves my symptoms instantly; 7 | 46
  Improves my breathing instantly; 1 | 14
  Improves my breathing instantly; 2 | 7
  Improves my breathing instantly; 3 | 10
  Improves my breathing instantly; 4 | 9
  Improves my breathing instantly; 5 | 16
  Improves my breathing instantly; 6 | 31
  Improves my breathing instantly; 7 | 46
  Works as good as medicated nasal sprays; 1 | 21
  Works as good as medicated nasal sprays; 2 | 6
  Works as good as medicated nasal sprays; 3 | 10
  Works as good as medicated nasal sprays; 4 | 6
  Works as good as medicated nasal sprays; 5 | 15
  Works as good as medicated nasal sprays; 6 | 23
  Works as good as medicated nasal sprays; 7 | 52
  Works better than medicated nasal sprays; 1 | 23
  Works better than medicated nasal sprays; 2 | 5
  Works better than medicated nasal sprays; 3 | 10
  Works better than medicated nasal sprays; 4 | 6
  Works better than medicated nasal sprays; 5 | 15
  Works better than medicated nasal sprays; 6 | 26
  Works better than medicated nasal sprays; 7 | 48

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the investigational product, and until 3 days following last administration of the investigational product.
Arm/Group | CO2 Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 75/147
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CO2 Nasal Spray (N=147)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 37 (75)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 12 (22)
Headache (Nervous system disorders) | 10 (10)
Application site pain (General disorders) | 9 (18)
Medical device site reaction (General disorders) | 3 (4)
Lacrimation increased (Eye disorders) | 11 (18)
Abdominal distension (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.